CLINICAL TRIAL: NCT07290231
Title: Effects of Core Strengthening Exercises With Diapgragmatic Breathing Versus Core Strengthening Exercises With Pilate Breathing in Diabetes Type II Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/93
Record Dates: First submitted 2025-09-11; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Type II
Keywords: core strengthening exercises; Pilate breathing exercises; diaphragmatic breathing exercises; Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be kept blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core strengthening with diaphragmatic breathing (Experimental): detailed components of core strengthening exercises and diaphragmatic breathing
  Interventions: Other: Core Strengthening with Diaphragmatic Breathing
- core strengthening with pilate breathing (Experimental): detailed components of core strengthening exercises and pilate breathing
  Interventions: Other: core strengthening with pilate breathing

INTERVENTIONS:
Other: Core Strengthening with Diaphragmatic Breathing — Swiss Ball Seated Marching: Sit on the ball with feet flat on the floor, hip-width apart. Keep the back straight and core engaged. Slowly lift right foot a few inches off the ground. Hold for 1-2 seconds, then lower. Lift left foot the same way. Continue alternating in a slow, controlled motion.
  Arms: core strengthening with diaphragmatic breathing
Other: core strengthening with pilate breathing — Pilates Breathing Sit/lie in neutral spine, hand on ribs & stomach. Inhale through nose, expand ribs (not shoulders). Exhale, draw navel to spine, engage core. Core Strengthening Abdominal Bracing: Tighten abs, hold while breathing. Pelvic Tilt: Flatten lower back, lift tailbone slightly. Hold 5-10s. Dead Bug: Lower opposite arm & leg, return. Alternate. Quadruped (Bird Dog): On all fours, extend opposite arm & leg. Hold 2-3s. Plank: Forearms down, straight body. Hold 20-60s. Bridge: Lift hips, squeeze glutes, lower slowly. Segmental Rolling: Roll with upper body first, then lower body. Swiss Ball Marching: Sit tall, lift one foot at a time.
  Arms: core strengthening with pilate breathing

SUMMARY:
Diabetes type II is a metabolic syndrome involving high sugar levels known as hyperglycemia. It can impair pulmonary function through reduced lung elasticity and gas exchange and weaken core muscles due to inflammation and muscle atrophy. Literature has shown the individual effects of these exercises on quality of life. However, no study has yet evaluated the combined effects of these exercises on different variables such as lung function, functional capacity, and blood sugar levels.

OBJECTIVE: The objective of this study is to compare the effects of diaphragmatic breathing and Pilates breathing, combined with core strengthening exercises, on lung function, functional capacity, blood sugar levels, and quality of life. The study aims to determine which breathing technique provides greater physiological and functional benefits.

METHOD: The study will be a Randomized control trial consisting of two groups subjects meeting the inclusion criteria will be selected for the study. The subjects will then be randomly assigned to two groups. One group will receive Diaphragmatic breathing with core strengthening exercises and other group will receive Pilate breathing with core strengthening exercises. Before initiating the treatment procedure following would be assessed for all the patients: Pulmonary Function, Functional Capacity, Blood sugar levels and quality of life. Afterwards a treatment regime distributed over the course of six weeks will be given to all patients. After the interventions Pulmonary function, Functional capacity, Blood sugar levels and Quality of life would be reassessed. Data would be analyzed to evaluate the outcomes.

DATA COLLECTION PROCEDURE: The participants eligible for the study according to inclusion and exclusion criteria would be recruited for the study voluntarily and referred from Medical OPD of Fauji Foundation Hospital and Rehab OPD of Fauji Foundation Hospital. The purpose of this study along with the treatment plan would be explained to the participants in the language they understand their best and informed consent will be taken from the participants. A treatment regimen consisting of 18 weeks distributed over the course of six weeks will be provided to the patients in multidisciplinary lab of foundation University College of physical therapy

DETAILED DESCRIPTION:
Diabetes type II is an expanding global problem linked to several factors such as obesity, unhealthy diet, and physical inactivity. The two most common causes are impaired insulin secretion or insulin resistance. Diabetes type II is a major health burden for the elderly population, affecting approximately 25% of individuals over the age of 65 years. Recently, increased attention has been paid to the loss of muscle power and sarcopenia in individuals with type II diabetes, as these conditions compromise both physical and psychological health, significantly affecting overall quality of life. Diabetes type II is a heterogeneous disorder affecting multiple organs. The alveolar capillary network, a large microvascular unit in the lungs, may be associated with the condition. Functional capacity is a strong predictor of survival in many diseases, including diabetes type II. Patients are more likely to experience functional impairments due to poor glycemic control and associated complications. Symptoms such as inadequate metabolic control, episodes of hypoglycemia, fear of hypoglycemia, and changes in lifestyle collectively lead to poor health-related quality of life, with reductions in functional performance. Activities of daily living and overall quality of life are often most affected by vascular complications in diabetes type II. Reduced lung function and impaired gas transfer are also linked to the disease. Chronic hyperglycemia causes the production of reactive oxygen species due to a process known as non-protein enzymatic glycation. Advanced glycation and continuous oxidative stress trigger a chronic inflammatory response. Additionally, there is a considerable decrease in glucose uptake in the skeletal muscles of patients with diabetes type II. Due to impaired insulin production and utilization, patients experience a constant state of elevated blood sugar levels that can lead to severe short-term and long-term consequences. Diabetes type II, therefore, represents a complex disorder characterized by defects in insulin production and utilization. Research also indicates that diets containing high sugar content, refined foods, and high-calorie foods significantly increase the risk of developing diabetes type II.

This study aims to explore the combined effects of treatment regimens on pulmonary function, functional capacity, random blood sugar levels, and quality of life. The investigation seeks to provide a deeper understanding of the effects of these interventions on various health variables.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed patients with Type II diabetes confirmed by a medical specialist, general practitioner, or endocrinologist from FFH or private hospital settings in Rawalpindi and Islamabad.
* Age between 30 and 55 years.
* Both male and female patients.
* Willingness to participate in the exercise program and ability to provide informed consent.
* On a stable regimen of anti-diabetic medications for at least three months prior to the study.

Exclusion Criteria:

* Patients with Type I diabetes, diabetes insipidus, or gestational diabetes.
* Diagnosed chronic respiratory diseases such as COPD or asthma unrelated to diabetes.
* History of any abdominal, orthopedic, or spinal surgery that could interfere with balance.
* Uncontrolled cardiovascular conditions such as arrhythmias or recent myocardial infarction.
* Morbid obesity (BMI > 40).
* Pregnant women.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
pulmonary Function | 6 weeks
  Pulmonary function will be assessed using spirometry following standard ATS/ERS procedures. Key parameters recorded will include FVC, FEV₁, and the FEV₁/FVC ratio. Spirometry will be used to evaluate baseline respiratory status and monitor any changes over time.
Functional capacity | 6 weeks
  Functional capacity will be assessed using the 6-Minute Walk Test (6MWT). Participants will be instructed to walk at their usual pace for six minutes along a standardized, measured corridor. The total distance walked (in meters) will be recorded as the outcome. Standardized encouragement and safety monitoring will be followed according to established guidelines.
Blood sugar levels | 6 weeks
  Blood sugar level will be measured using a calibrated glucometer. A capillary blood sample will be obtained via finger-prick, and glucose concentration will be recorded in mg/dL according to standard operating procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, 44000, Islamabad, Pakistan